CLINICAL TRIAL: NCT01671215
Title: Endometrial and Myometrial Changes, With and Without Fibroids
Status: Withdrawn | Type: Observational
Why Stopped: no enrollment
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC120026CTIL
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2012-04

CONDITIONS: Fibroids
Keywords: endometrium; myometrium; fibroids; uterine malformations
MeSH Terms: conditions — Leiomyoma; Uterine Anomalies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
fibroids are common among women in fertile age. the relation between fibroids and infertility is controversial. our goal is to claculate a ratio between uterine cavity - endometrium & myometrium in normal uterine s and study the interference of the cavity in uterine s with fibroids.

DETAILED DESCRIPTION:
phase 1-

1. retrospective measurments of uterine dimensions of 100 women with normal uterin
2. measurment of the above during different sycle days in the same woman. 30 women.

phase 2- retrospective measurments of 500 uterine dimensions of women with fibroids phase 3- the same for 400 uterine malformations

ELIGIBILITY:
Inclusion Criteria:

* women at IVF unit

Exclusion Criteria:

* inabilty to measure propperly the uterine dimensions

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women at the age of 20-45
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
ratio between normal & abnormal(by fibroid) uterine cavity | year

SECONDARY OUTCOMES:
ratio between endometriom & myometrium area, circumference &n volume | year

CONTACTS AND LOCATIONS:
Overall Officials: ronni tepper, md, Principal Investigator — Tel Aviv University
Locations (1):
- Meir medical center, Kfar Saba, Israel